CLINICAL TRIAL: NCT04587453
Title: A Randomised, Double-blind, Placebo-controlled, Phase 3 Trial to Evaluate the Efficacy and Safety of Tralokinumab in Combination With Topical Corticosteroids in Japanese Subjects With Moderate-to-severe Atopic Dermatitis Who Are Candidates for Systemic Therapy
Brief Title: Tralokinumab in Combination With Topical Corticosteroids in Japanese Subjects With Moderate-to-severe Atopic Dermatitis
Acronym: ECZTRA 8
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0162-1343
Record Dates: First submitted 2020-09-29; First posted 2020-10-14 (Actual); Results first posted 2022-09-22 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2022-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — tralokinumab; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Neither the trial participant nor any of the investigator or LEO pharma staff who are involved in the treatment or clinical evaluation and monitoring of the participants will be aware of the treatment received. The packaging and labelling of the investigational medicinal product (IMP) will contain no evidence of their identity. Since tralokinumab and placebo are visually distinct and not matched for viscosity, IMP will be handled and administered by a qualified, unblinded healthcare professional at the site who will not be involved in the management of trial participants and who will not perform any of the assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tralokinumab+TCS (Experimental): Week 0 to Week 16: Tralokinumab will be given as subcutaneous injections. Participants will receive tralokinumab loading dose on Day 0 followed by multiple tralokinumab injections. The last administration will occur at Week 14. Topical corticosteroids (TCS) will be administered as needed.
  Interventions: Drug: Tralokinumab; Other: Topical corticosteroids (TCS)
- Placebo+TCS (Placebo Comparator): Week 0 to Week 16: Placebo will be given as subcutaneous injections. Participants will receive placebo loading dose on Day 0 followed by multiple placebo injections. The last administration will occur at Week 14. Topical corticosteroids (TCS) will be administered as needed.
  Interventions: Drug: Placebo; Other: Topical corticosteroids (TCS)

INTERVENTIONS:
Drug: Tralokinumab — Tralokinumab is a human recombinant monoclonal antibody of the immunoglobulin G4 subclass that specifically binds to human interleukin-13 (IL-13) and blocks the interaction with IL-13 receptors. It is presented as a liquid formulation for subcutaneous administration.
  Arms: Tralokinumab+TCS
Drug: Placebo — Placebo contains the same excipients in the same concentration only lacking tralokinumab.
  Arms: Placebo+TCS
Other: Topical corticosteroids (TCS) — TCS administered as needed.

SUMMARY:
Primary objective:

To evaluate the efficacy of tralokinumab in combination with topical corticosteroids (TCS) compared with placebo in combination with TCS in treating moderate-to-severe atopic dermatitis (AD).

Secondary objectives:

To evaluate the efficacy of tralokinumab in combination with TCS on severity and extent of AD, itch, health-related quality of life, and health care resource utilisation compared with placebo in combination with TCS.

To assess the safety of tralokinumab in combination with TCS when used to treat moderate-to-severe AD for 16 weeks.

ELIGIBILITY:
Key inclusion criteria:

* Japanese subject aged 18 years and above.
* Diagnosis of AD as defined by the Hanifin and Rajka (1980) criteria for AD.
* History of AD for 1 year or more.
* A recent history (within 1 year before screening) of inadequate response to treatment with topical medication.
* AD involvement of 10% or more body surface area at screening and at baseline according to component A of SCORAD.
* Applied a stable dose of emollient twice daily (or more, as needed) for at least 14 days before randomisation.

Key exclusion criteria:

* Subjects for whom TCS are medically inadvisable e.g. due to important side effects or safety risks in the opinion of the investigator.
* Active dermatologic conditions that may confound the diagnosis of AD or would interfere with assessment of treatment.
* Use of tanning beds or phototherapy within 6 weeks prior to randomisation.
* Treatment with systemic immunosuppressive/immunomodulating drugs and/or systemic corticosteroids within 4 weeks prior to randomisation.
* Treatment with TCS, topical calcineurin inhibitors, topical phosphodiesterase-4 inhibitors, or topical Janus kinase inhibitors within 2 weeks prior to randomisation.
* Receipt of any marketed biological therapy (i.e. immunoglobulin, anti-immunoglobulin E) including dupilumab or investigational biologic agents 3 to 6 months prior to randomisation.
* Active skin infections within 1 week prior to randomisation.
* Clinically significant infection within 4 weeks prior to randomisation.
* A helminth parasitic infection within 6 months prior to the date informed consent is obtained.
* Tuberculosis requiring treatment within the 12 months prior to screening.
* Known primary immunodeficiency disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (22):
- Japan (22):
  - LEO Investigational Site, Nagoya, Aichi-ken
  - LEO Investigational Site, Ichikawa, Chiba
  - LEO Investigational Site, Ichikawa-shi, Chiba
  - LEO Investigational Site, Chikushino-shi, Fukuoka
  - LEO Investigational Site, Asahikawa, Hokkaido
  - LEO Investigational Site, Chuo-Ku-Sapporo, Hokkaido
  - LEO Investigational Site, Obihiro-shi, Hokkaido
  - LEO Investigational Site, Sapporo, Hokkaido
  - LEO Investigational Site, Nishinomiya, Hyōgo
  - LEO Investigational Site, Nonoichi, Ishikawa-ken
  - LEO Investigational Site, Kagoshima, Kagoshima-ken
  - LEO Investigational Site, Kawasaki-shi, Kanagawa
  - LEO Investigational Site, Yokohama, Kanagawa
  - LEO Investigational Site, Kamigyō-ku, Kyoto
  - LEO Investigational Site, Tokyo, Minato
  - LEO Investigational Site, Osaka, Osaka
  - LEO Investigational Site, Sakai-shi, Osaka
  - LEO Investigational Site, Toyonaka-shi, Osaka
  - LEO Investigational Site, Koto-ku, Tokyo
  - LEO Investigational Site, Setagaya City, Tokyo
  - LEO Investigational Site, Shinjuku-ku, Tokyo
  - LEO Investigational Site, Fukuoka

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject first visit: 27-Oct-2020. Subjects were recruited at 25 sites in Japan.
Pre-assignment Details: 126 subjects were screened. 20 subjects were screening failures. 106 subjects were included in the trial and randomised 1:1 to tralokinumab+TCS and placebo+TCS.
  All randomised subjects received at least 1 dose of investigational medicinal product (IMP).
Groups:
- Tralokinumab+TCS: Treatment period (Week 0 to Week 16): Participants received 600 mg tralokinumab (4 subcutaneous injections) as a loading dose on Day 0. Then they received 300 mg tralokinumab (2 subcutaneous injections) every 2 weeks until Week 14. Topical corticosteroids (TCS) (mometasone furoate, 0.1% cream, Japan classification: Very strong) were applied on the skin as needed.
  Safety follow-up period (Week 17 to Week 20): Period without treatment.
  Tralokinumab is a human recombinant monoclonal antibody of the immunoglobulin G4 subclass that specifically binds to human interleukin-13 (IL-13) and blocks the interaction with IL-13 receptors. It is presented as a liquid formulation for subcutaneous administration.
- Placebo+TCS: Treatment period (Week 0 to Week 16): Participants received 4 subcutaneous injections of placebo (resembling a loading dose) on Day 0. Then they received 2 subcutaneous injections of placebo every 2 weeks until Week 14. Topical corticosteroids (TCS) (mometasone furoate, 0.1% cream, Japan classification: Very strong) were applied on the skin as needed.
  Safety follow-up period (Week 17 to Week 20): Period without treatment.
  Placebo contains the same excipients in the same concentration, but without the active ingredient of tralokinumab.
Period: Treatment Period (Week 0 to Week 16)
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Started | 53 | 53
Full Analysis Set (All participants randomised and exposed to IMP.) | 53 | 53
Safety Analysis Set (All participants exposed to IMP.) | 53 | 53
Completed (Participants attended the Week 16 visit (end of treatment visit).) | 53 | 52
Not Completed | 0 | 1
Not completed — Premature (before Week 16) discontinuation of IMP | 0 | 1
Period: Safety Follow-up (Week 16 to Week 20)
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Started (Date of last contact was after the date of exposure end.) | 8 | 3
Not Started (Transferred to the long-term extension trial ECZTEND (LP0162-1337) instead of entering the safety follow-up period.) | 45 | 49
Safety Follow-up Analysis Set (Date of last contact was after the date of exposure end.) | 8 | 4 (1 subject prematurely discontinued treatment before Week 16, but did have contact after last exposure date and was therefore included in the safety follow-up analysis set.)
Completed (Completed the safety follow-up period with a safety follow-up visit.) | 8 (1 participant transferred to ECZTEND (LP0162-1337) at the safety follow-up visit.) | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomised subjects
Groups:
- Tralokinumab+TCS: Treatment period (Week 0 to Week 16): Participants were treated with 300 mg tralokinumab every 2 weeks until Week 14, after a loading dose of 600 mg tralokinumab at Week 0. TCS was applied on the skin as needed.
- Placebo+TCS: Treatment period (Week 0 to Week 16): Participants received placebo every 2 weeks until Week 14, after a loading dose of placebo at Week 0. TCS was applied on the skin as needed.
- Total: Total of all reporting groups
Arm/Group | Tralokinumab+TCS | Placebo+TCS | Total
Number analyzed (Participants) | 53 | 53 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 53 | 105
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (13.7) | 38.9 (12.1) | 39.0 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 22 | 39
  Male | 36 | 31 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 53 | 53 | 106
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 53 | 53 | 106
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 53 | 53 | 106
Age at onset of atopic dermatitis [Median (Inter-Quartile Range); unit: years] | 3.0 [1.0 to 6.0] | 5.0 [1.0 to 14.0] | 4.0 [1.0 to 10.0]
Duration of atopic dermatitis [Mean (Standard Deviation); unit: years] | 32.0 (13.0) | 30.8 (14.0) | 31.4 (13.5)
Body surface area (BSA) with atopic dermatitis [Mean (Standard Deviation); unit: percentage of BSA affected] | 66.6 (20.7) | 64.4 (18.5) | 65.5 (19.6)
Investigator's Global Assessment (IGA) [Count of Participants; unit: Participants] — IGA is an instrument used in clinical trials to rate the severity of the participant's global AD and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
  Participants
    Clear | 0 | 0 | 0
    Almost clear | 0 | 0 | 0
    Mild | 0 | 0 | 0
    Moderate | 23 | 23 | 46
    Severe | 30 | 30 | 60
Eczema Area and Severity Index (EASI) score [Mean (Standard Deviation); unit: score on a scale] — EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. EASI is a composite index with scores ranging from 0 to 72, where higher values indicate a more severe or more extensive condition.
  score on a scale | 37.12 (15.71) | 32.30 (12.32) | 34.71 (14.25)
Scoring Atopic Dermatitis (SCORAD) [Mean (Standard Deviation); unit: score on a scale] — SCORAD is calculated as A/5+7B/2+C (max total score = 103, with higher values indicating more severe disease): A) Extent of AD lesions (sum of % of all defined body areas; max score = 100%); B) Severity of AD lesions (6 specific symptoms assessed on a representative area using the scale: 0 = none/absent, 1 = mild, 2 = moderate, 3 = severe; max score = 18); C) Subjective symptoms (subjective assessment of itch and sleeplessness over the last 3 days/nights for each symptom on a VAS scale: 0 = no itch or trouble sleeping, 10 = unbearable itch or a lot of trouble sleeping; max score = 20).
  score on a scale | 71.72 (13.79) | 69.82 (12.39) | 70.77 (13.08)
Dermatology Life Quality Index (DLQI) [Mean (Standard Deviation); unit: score on a scale] — DLQI consists of 10 items addressing the participant's perception of the impact of their skin disease on different aspects of their health-related quality of life over the past week, such as dermatology-related symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the treatment. Each item is scored on a 4-point Likert scale (0=not at all ⁄ not relevant; 1=a little; 2=a lot; 3=very much). The total score is the sum of the 10 items (ranging from 0 to 30), with higher scores indicating poorer health-related quality of life.
  score on a scale | 13.09 (6.92) | 14.30 (6.39) | 13.70 (6.65)
Worst Daily Pruritus numeric rating scale (NRS) [Mean (Standard Deviation); unit: score on a scale] — Participants assess their worst itch severity over the past 24 hours using an 11-point NRS (Worst Daily Pruritus NRS) with 0 indicating 'no itch' and 10 indicating 'worst itch imaginable'.
  score on a scale | 7.60 (1.65) | 7.81 (1.37) | 7.71 (1.51)

OUTCOME MEASURES:

1. Primary Outcome: Investigator's Global Assessment (IGA) Score of 0 (Clear) or 1 (Almost Clear) at Week 16
Description: IGA is an instrument used in clinical trials to rate the severity of the participant's global AD and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Time Frame: Week 16
Population: Full analysis set: 106 subjects, all randomised and treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 53 | 53
Participants | 17 | 14
Statistical Analysis 1: Comparison: Tralokinumab+TCS vs Placebo+TCS; Responders were considered those meeting an IGA score of 0 or 1 (clear or almost clear). Subjects with missing data or subjects who had received rescue medication prior to Week 16 were considered non-responders in the primary analysis of the primary estimand; Test type: Other — No formal testing was performed. Confidence intervals (CIs) are presented with two sided 95% degree of confidence; Risk Difference (RD) = 5.7, 95% CI 2-sided [-11.2 to 22.5] — Mantel-Haenzel risk difference, stratified by baseline IGA

2. Primary Outcome: At Least 75% Reduction in Eczema Area and Severity Index (EASI75) at Week 16
Description: Eczema Area and Severity Index (EASI) is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. EASI is a composite index with scores ranging from 0 to 72, where higher values indicate a more severe or more extensive condition.
Time Frame: Week 0 to Week 16
Population: Full analysis set: 106 subjects, all randomised and treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 53 | 53
Participants | 38 | 30
Statistical Analysis 1: Comparison: Tralokinumab+TCS vs Placebo+TCS; Subjects with 75% reduction in EASI were considered responders. Subjects with missing data or subjects who had received rescue medication prior to Week 16 were considered non-responders in the primary analysis of the primary estimand; Test type: Other — No formal testing was performed. CIs are presented with two sided 95% degree of confidence; Risk Difference (RD) = 15.1, 95% CI 2-sided [-2.9 to 33.0] — Mantel-Haenzel risk difference, stratified by baseline IGA

3. Secondary Outcome: Change in Scoring Atopic Dermatitis (SCORAD) Total Score From Baseline to Week 16
Description: SCORAD is a validated tool to evaluate the AD disease based on 3 components:
  * A) The extent of AD lesions. Assessed as percentage of each defined body area and reported as sum of all areas (max score = 100%).
  * B) The severity of AD lesions. The intensity of 6 specific symptoms on a representative area was assessed using the scale: 0 = none/absent, 1 = mild, 2 = moderate, 3 = severe (max score = 18).
  * C) Subjective symptoms. The itch and sleeplessness over the last 3 days/nights was recorded for each symptom by the subject on a VAS scale: 0 = no itch or trouble sleeping, 10 = unbearable itch or a lot of trouble sleeping (max score = 20).
  The SCORAD was calculated as: A/5+7B/2+C. The maximum total score is 103, with higher values indicating more severe disease.
Time Frame: Week 0 to Week 16
Population: Full analysis set: 106 subjects, all randomised and treated.
Measure: Least Squares Mean (Standard Error); unit: change in score on a scale
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 53 | 53
change in score on a scale | -44.1 (2.61) | -39.0 (2.61)
Statistical Analysis 1: Comparison: Tralokinumab+TCS vs Placebo+TCS; Test type: Other — No formal testing was performed. CIs are presented with two sided 95% degree of confidence; Mean Difference (Net) = -5.1, 95% CI 2-sided [-12.4 to 2.3] — Analysis of covariance (ANCOVA). Worst observation carried forward for all subjects who prior to Week 16 had received rescue medication. Multiple imputation of missing values for subjects who had not received rescue medication

4. Secondary Outcome: Change in Dermatology Life Quality Index (DLQI) Score From Baseline to Week 16.
Description: DLQI consists of 10 items addressing the participant's perception of the impact of their skin disease on different aspects of their health-related quality of life over the past week, such as dermatology-related symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the treatment. Each item is scored on a 4-point Likert scale (0=not at all ⁄ not relevant; 1=a little; 2=a lot; 3=very much). The total score is the sum of the 10 items (ranging from 0 to 30), with higher scores indicating poorer health-related quality of life.
Time Frame: Week 0 to Week 16
Population: Full analysis set: 106 subjects, all randomised and treated.
Measure: Least Squares Mean (Standard Error); unit: change in score on a scale
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 53 | 53
change in score on a scale | -10.0 (0.56) | -8.8 (0.56)
Statistical Analysis 1: Comparison: Tralokinumab+TCS vs Placebo+TCS; Test type: Other — No formal testing was performed. CIs are presented with two sided 95% degree of confidence; Mean Difference (Net) = -1.1, 95% CI 2-sided [-2.7 to 0.5] — ANCOVA. Worst observation carried forward for all subjects who prior to Week 16 had received rescue medication. Multiple imputation of missing values for subjects who had not received rescue medication

5. Secondary Outcome: Reduction of Worst Daily Pruritus Numeric Rating Scale (NRS) Score (Weekly Average) of at Least 4 From Baseline to Week 16
Description: Participants assessed the itch for the past 24 hours using the Worst Daily Pruritus NRS, consisting of 11 points, with 0 indicating 'no itch' and 10 indicating 'worst itch imaginable'.
Time Frame: Week 0 to Week 16
Population: Full analysis set: 106 subjects, all randomised and treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 53 | 53
Participants | 34 | 36
Statistical Analysis 1: Comparison: Tralokinumab+TCS vs Placebo+TCS; Subjects with at least a reduction of 4 in the worst daily pruritus NRS score were considered responders. Subjects who had received rescue medication were considered non-responders. Subjects with missing data at Week 16 were imputed as non-responders; Test type: Other — No formal testing was performed. CIs are presented with two sided 95% degree of confidence; Risk Difference (RD) = -3.8, 95% CI 2-sided [-21.7 to 14.2] — Mantel-Haenszel risk difference, stratified by baseline IGA

6. Secondary Outcome: At Least 90% Reduction in EASI (EASI90) at Week 16
Description: EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. EASI is a composite index with scores ranging from 0 to 72, where higher values indicate a more severe or more extensive condition.
Time Frame: Week 0 to Week 16
Population: Full analysis set: 106 subjects, all randomised and treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 53 | 53
Participants | 24 | 16
Statistical Analysis 1: Comparison: Tralokinumab+TCS vs Placebo+TCS; Subjects with a reduction of 90% in EASI were considered responders. Subjects who had received rescue medication were considered non-responders. Subjects with missing data were imputed as non-responders; Test type: Other — No formal testing was performed. CIs are presented with two sided 95% degree of confidence; Risk Difference (RD) = 15.1, 95% CI 2-sided [-3.0 to 33.2] — Mantel-Haenszel risk difference, stratified by baseline IGA

7. Secondary Outcome: At Least 50% Reduction in EASI (EASI50) at Week 16
Description: as for outcome 6
Time Frame: Week 0 to Week 16
Population: Full analysis set: 106 subjects, all randomised and treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 53 | 53
Participants | 45 | 42
Statistical Analysis 1: Comparison: Tralokinumab+TCS vs Placebo+TCS; Subjects with at least 50% reduction in EASI were considered responders. Subjects who had received rescue medication were considered non-responders. Subjects with missing data were imputed as non-responders; Test type: Other — No formal testing was performed. CIs are presented with two sided 95% degree of confidence; Risk Difference (RD) = 5.7, 95% CI 2-sided [-9.0 to 20.3] — Mantel-Haenszel risk difference, stratified by baseline IGA

8. Secondary Outcome: Percentage Change in EASI Score From Baseline to Week 16
Description: as for outcome 6
Time Frame: Week 0 to Week 16
Population: Full analysis set: 106 subjects, all randomised and treated.
Measure: Least Squares Mean (Standard Error); unit: percentage change in score on a scale
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 53 | 49
percentage change in score on a scale | -77.8 (3.70) | -73.5 (3.76)
Statistical Analysis 1: Comparison: Tralokinumab+TCS vs Placebo+TCS; Test type: Other — No formal testing was performed. CIs are presented with two sided 95% degree of confidence; Mean Difference (Net) = -4.3, 95% CI 2-sided [-14.9 to 6.3] — Repeated measurements Model: Change=Treatment*Week+Baseline*Week+Baseline IGA. Data after permanent discontinuation of IMP/initiation of rescue medication not included (4 subjects excluded). Week 2 change imputed as 0 if no post-baseline assessments

9. Secondary Outcome: Change in Worst Daily Pruritus NRS Score (Weekly Average) From Baseline to Week 16
Description: as for outcome 5
Time Frame: Week 0 to Week 16
Population: Full analysis set:106 subjects, all randomised and treated.
Measure: Least Squares Mean (Standard Error); unit: change in score on a scale
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 53 | 49
change in score on a scale | -4.6 (0.26) | -4.6 (0.27)
Statistical Analysis 1: Comparison: Tralokinumab+TCS vs Placebo+TCS; Test type: Other — No formal testing was performed. CIs are presented with two sided 95% degree of confidence; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.7 to 0.8] — [estimate comment as in outcome 8, analysis 1]

10. Secondary Outcome: Change in Eczema-related Sleep NRS Score (Weekly Average) From Baseline to Week 16
Description: Participants rated how much their eczema interfered with their sleep the last night using an 11-point NRS (0 indicating that it 'did not interfere' and 10 indicating that it 'completely interfered').
Time Frame: Week 0 to Week 16
Population: Full analysis set: 106 subjects, all randomised and treated.
Measure: Least Squares Mean (Standard Error); unit: change in score on a scale
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 53 | 49
change in score on a scale | -4.2 (0.25) | -4.1 (0.26)
Statistical Analysis 1: Comparison: Tralokinumab+TCS vs Placebo+TCS; Test type: Other — No formal testing was performed. CIs are presented with two sided 95% degree of confidence; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.9 to 0.6] — Repeated measurements model: Change=Treatment*Week+Baseline*Week+Baseline IGA. Data after permanent discontinuation of IMP/initiation of rescue medication not included (4 subjects excluded). Week 1 change imputed as 0 if no post-baseline assessments

11. Secondary Outcome: Change in Patient-Oriented Eczema Measure (POEM) Score Form Baseline to Week 16
Description: POEM consists of 7 items, each addressing a specific symptom (itching, sleep, bleeding, weeping, cracking, flaking, and dryness). Participants score how often they have experienced each symptom over the previous week, using a 5-point categorical response scale (0=no days; 1=1 to 2 days; 2=3 to 4 days; 3=5 to 6 days; 4=every day). The total score is the sum of the 7 items (ranging from 0 to 28) and reflects disease-related morbidity; higher scores indicate more severe disease.
Time Frame: Week 0 to Week 16
Population: Full analysis set: 106 subjects, all randomised and treated.
Measure: Least Squares Mean (Standard Error); unit: change in score on a scale
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 53 | 49
change in score on a scale | -14.4 (0.82) | -11.2 (0.83)
Statistical Analysis 1: Comparison: Tralokinumab+TCS vs Placebo+TCS; Test type: Other — No formal testing was performed. CIs are presented with two sided 95% degree of confidence; Mean Difference (Net) = -3.2, 95% CI 2-sided [-5.6 to -0.9] — [estimate comment as in outcome 8, analysis 1]

12. Secondary Outcome: Number of Treatment-emergent Adverse Events From Baseline to Week 16 Per Subject
Description: Number of events divided by patient years of exposure (= rate).
Time Frame: Week 0 to Week 16
Population: Safety analysis set: 106 subjects. Included all subjects exposed to IMP at least 1 time.
Measure: Number; unit: events per patient year of exposure
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 53 | 53
events per patient year of exposure | 605.9 | 332.8

13. Secondary Outcome: Number of Subjects With Presence of Treatment-emergent Anti-drug Antibodies (ADA) From Baseline to Week 16
Description: Anti-tralokinumab antibody levels were analyzed using a validated bioanalytical method. Positive treatment-emergent ADA was defined as ADA negative or missing at baseline, and at least one positive post-baseline ADA response. Negative treatment-emergent ADA was defined as ADA negative or missing at baseline, and all post-baseline ADA assessments negative.
Time Frame: Week 0 to Week 16
Population: Safety analysis set. Included all subjects exposed to IMP at least 1 time.
Measure: Number; unit: participants with treatment-emergent ADA
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 53 | 53
participants with treatment-emergent ADA | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment period: Week 0 to Week 16; Safety follow-up period: Week 16 to Week 20
Description: Safety analysis set: 106 subjects. Included all subjects exposed to IMP at least 1 time.
Groups:
- Treatment Period: Tralokinumab+TCS: During the treatment period (Week 0 to Week 16), participants were treated with 300 mg tralokinumab every 2 weeks until Week 14, after a loading dose of 600 mg tralokinumab at Week 0. TCS was applied on the skin as needed.
- Treatment Period: Placebo+TCS: During the treatment period (Week 0 to Week 16), participants received placebo every 2 weeks until Week 14, after a loading dose of placebo at Week 0. TCS was applied on the skin as needed.
- Safety Follow-up Period: Tralokinumab+TCS: No treatment was administered during the safety-follow-up period (Week 17 to Week 20). Participants received tralokinumab+TCS in the treatment period.
  Eligible participants were invited to enter a long-term extension trial conducted under a separate protocol (LP0162-1337, ECZTEND).
- Safety Follow-up Period: Placebo+TCS: No treatment was administered during the safety-follow-up period (Week 17 to Week 20). Participants received placebo+TCS in the treatment period.
  Eligible participants were invited to enter a long-term extension trial conducted under a separate protocol (LP0162-1337, ECZTEND).
Arm/Group | Treatment Period: Tralokinumab+TCS | Treatment Period: Placebo+TCS | Safety Follow-up Period: Tralokinumab+TCS | Safety Follow-up Period: Placebo+TCS
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/53 | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53 | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 28/53 | 19/53 | 2/8 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period: Tralokinumab+TCS (N=53) | Treatment Period: Placebo+TCS (N=53) | Safety Follow-up Period: Tralokinumab+TCS (N=8) | Safety Follow-up Period: Placebo+TCS (N=4)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 3 (12) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 5 (10) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (4) | 5 (6) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (3) | 1 (1) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 6 (7) | 4 (4) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial was not powered to show superiority of tralokinumab+TCS vs placebo+TCS, but to facilitate an evaluation of similarity with the treatment effect observed in the LP0162-1339 trial (EU and US). The first 16 weeks were similar in the 2 trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO Pharma A/S seeks publication of all clinical trials in peer-reviewed journals within 18 months after completion or termination of the clinical trial, regardless of whether the findings are positive or negative. If no publication is submitted by LEO Pharma A/S within these 18 months, the investigator has the right to publish the results from the clinical trial generated by him/herself.

DOCUMENTS (2):
  • Study Protocol (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT04587453/Prot_002.pdf
  • Statistical Analysis Plan (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT04587453/SAP_001.pdf